CLINICAL TRIAL: NCT04214951
Title: A Prospective Observational Study of Switching Eltrombopag and Recombinant Human Thrombopoietin In Primary Immune Thrombocytopenia
Brief Title: A Study of Eltrombopag and Recombinant Human Thrombopoietin In Primary Immune Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Clinical Professor, Peking University People's Hospital
Other Study IDs: ZXH-ITP2019
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Corticosteroid-resistant or Relapsed ITP
Keywords: Immune Thrombocytopenia; Recombinant human thrombopoietin; Eltrombopag; switching
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Thrombopoietin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recombinant human thrombopoietin (rh-TPO) group: Patients who fail previous steroids and eltrombopag and then switch to Rh-TPO will be enrolled. The reason for switch will be recorded. Patients will be given rh-TPO 300 U/kg once daily for 21 days. Rh-TPO will be terminated any time the platelet counts increased above 100 × 10^9/L. The efficacy, safety, and patient/physician preference will be assessed.
  Interventions: Drug: Recombinant human thrombopoietin (rh-TPO)
- Eltrombopag group: Patients who fail previous steroids and rh-TPO and then switch to eltrombopag will be enrolled. The reason for switch will be recorded. Patients will be given eltrombopag 50mg once daily for 6 weeks. Eltrombopag will be terminated any time the platelet counts increased above 300× 10^9/L.The efficacy, safety, and patient/physician preference will be assessed.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Patients will be given eltrombopag 50mg once daily for 6 weeks.
  Groups: Eltrombopag group
Drug: Recombinant human thrombopoietin (rh-TPO) — Patients will be given rh-TPO 300 U/kg once daily for 21 days.
  Groups: Recombinant human thrombopoietin (rh-TPO) group

SUMMARY:
Thrombopoietin Receptor Agonists (TPO-ra) are novel treatments for patients with refractory Primary Immune Thrombocytopenia (ITP). Rh-TPO and eltrombopag increase the number of platelets through different mechanism. If there is cross-resistance between 2 drugs for the treatment of adult ITP is still no answer. The purpose of this study is to investigate the efficacy and safety of switching eltrombopag and Rh-TPO in adults with ITP.

DETAILED DESCRIPTION:
Non-interventional study. Patients who fail previous steroids and receive rh-TPO and then switch to EPAG or vice versa will be enrolled. The reason for switch will be recorded. Patients in the rh-TPO group were given rh-TPO 300 U/kg once daily for 21 days, and those in the eltrombopag group were given eltrombopag 50mg once daily for 6 weeks. Rh-TPO and eltrombopag were terminated any time the platelet counts increased above 100 × 10^9/L in the rh-TPO group and 300 × 10^9/L in the eltrombopag group. The efficacy, safety, and patient/physician preference will be assessed and compared between the two agents.

ELIGIBILITY:
Inclusion Criteria:

1.18 years or older

2.Primary ITP

3.Platelet count ≤ 30 × 109/l

4.Normal neutrophils, reticulocyte count, creatinine and liver enzyme values

5.Available follow-up of 2 months at least for each period

6.Failed initial glucocorticosteroid treatment

7.Unwillingness to accept splenectomy or failed splenectomy

-

Exclusion Criteria:

1. HIV, hepatitis B or C, Helicobacter pylori infection
2. Malignancy
3. Congenital or acquired immunologic deficit
4. History of thrombosis plus two or more risk factors
5. Nursing or pregnant women
6. Abnormal liver and renal functions: AST/ALT/total bilirubin ≥1.5 × ULN, creatinine ≥1.5 mg/dl
7. Severe heart and lung dysfunctions -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ITP patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Hui Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neunert C, Lim W, Crowther M, Cohen A, Solberg L Jr, Crowther MA; American Society of Hematology. The American Society of Hematology 2011 evidence-based practice guideline for immune thrombocytopenia. Blood. 2011 Apr 21;117(16):4190-207. doi: 10.1182/blood-2010-08-302984. Epub 2011 Feb 16. PMID 21325604
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Ghanima W, Godeau B, Cines DB, Bussel JB. How I treat immune thrombocytopenia: the choice between splenectomy or a medical therapy as a second-line treatment. Blood. 2012 Aug 2;120(5):960-9. doi: 10.1182/blood-2011-12-309153. Epub 2012 Jun 26. PMID 22740443
- [Background] Deutsch VR, Tomer A. Advances in megakaryocytopoiesis and thrombopoiesis: from bench to bedside. Br J Haematol. 2013 Jun;161(6):778-93. doi: 10.1111/bjh.12328. Epub 2013 Apr 18. PMID 23594368
- [Background] Kuter DJ. The biology of thrombopoietin and thrombopoietin receptor agonists. Int J Hematol. 2013 Jul;98(1):10-23. doi: 10.1007/s12185-013-1382-0. Epub 2013 Jul 3. PMID 23821332
- [Background] Bussel JB, Lakkaraja M. Thrombopoietic agents: there is still much to learn. Presse Med. 2014 Apr;43(4 Pt 2):e69-78. doi: 10.1016/j.lpm.2014.02.008. Epub 2014 Mar 27. PMID 24680422
- [Background] Wormann B. Clinical indications for thrombopoietin and thrombopoietin-receptor agonists. Transfus Med Hemother. 2013 Oct;40(5):319-25. doi: 10.1159/000355006. Epub 2013 Sep 11. PMID 24273485
- [Background] Wang S, Yang R, Zou P, Hou M, Wu D, Shen Z, Lu X, Li Y, Chen X, Niu T, Sun H, Yu L, Wang Z, Zhang Y, Chang N, Zhang G, Zhao Y. A multicenter randomized controlled trial of recombinant human thrombopoietin treatment in patients with primary immune thrombocytopenia. Int J Hematol. 2012 Aug;96(2):222-8. doi: 10.1007/s12185-012-1124-8. Epub 2012 Jun 30. PMID 22753022
- [Background] Erickson-Miller CL, Delorme E, Tian SS, Hopson CB, Landis AJ, Valoret EI, Sellers TS, Rosen J, Miller SG, Luengo JI, Duffy KJ, Jenkins JM. Preclinical activity of eltrombopag (SB-497115), an oral, nonpeptide thrombopoietin receptor agonist. Stem Cells. 2009 Feb;27(2):424-30. doi: 10.1634/stemcells.2008-0366. PMID 19038790
- [Background] Erhardt JA, Erickson-Miller CL, Aivado M, Abboud M, Pillarisetti K, Toomey JR. Comparative analyses of the small molecule thrombopoietin receptor agonist eltrombopag and thrombopoietin on in vitro platelet function. Exp Hematol. 2009 Sep;37(9):1030-7. doi: 10.1016/j.exphem.2009.06.011. Epub 2009 Jul 24. PMID 19631713
- [Background] Gonzalez-Porras JR, Godeau B, Carpenedo M. Switching thrombopoietin receptor agonist treatments in patients with primary immune thrombocytopenia. Ther Adv Hematol. 2019 May 9;10:2040620719837906. doi: 10.1177/2040620719837906. eCollection 2019. PMID 31156798
- [Background] Cantoni S, Carpenedo M, Mazzucconi MG, De Stefano V, Carrai V, Ruggeri M, Specchia G, Vianelli N, Pane F, Consoli U, Artoni A, Zaja F, D'adda M, Visentin A, Ferrara F, Barcellini W, Caramazza D, Baldacci E, Rossi E, Ricco A, Ciminello A, Rodeghiero F, Nichelatti M, Cairoli R. Alternate use of thrombopoietin receptor agonists in adult primary immune thrombocytopenia patients: A retrospective collaborative survey from Italian hematology centers. Am J Hematol. 2018 Jan;93(1):58-64. doi: 10.1002/ajh.24935. Epub 2017 Nov 9. PMID 28983953
- [Derived] Cai X, Fu H, Zhao X, Lu J, Jiang Q, Chang Y, Huang X, Zhang X. Switching between eltrombopag and recombinant human thrombopoietin in patients with immune thrombocytopenia: an observational study. Chin Med J (Engl). 2022 Oct 5;135(19):2344-2350. doi: 10.1097/CM9.0000000000002346. PMID 36535011

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Started | 50 | 50
Completed | 10 | 10
Not Completed | 40 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Thrombopoietin (Rh-TPO) Group | Eltrombopag Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [19 to 45] | 28 [18 to 39] | 29 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at 6 Weeks After Switching
Description: The percentage of patients who have reached platelet count ≥ 50×10^9/L at 6 weeks after switching.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

2. Secondary Outcome: Treatments Associated Adverse Events
Description: Adverse event/serious adverse event associated with study drugs during 6 weeks after switching
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
participants | 3 | 1

3. Secondary Outcome: Reasons of Switching
Description: Reasons of switching eltrombopag and rh-TPO will be recorded, including lack of efficacy, patient preference, side effects, platelet count fluctuation
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
Participants
  lack of efficacy | 2 | 2
  patient preference | 5 | 1
  side effects | 3 | 5
  platelet count fluctuation | 0 | 2

4. Secondary Outcome: Number of Participants With Bleeding Events
Description: Number of participants with bleeding events of the two groups during 6 weeks after switching
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
Participants | 2 | 4

5. Secondary Outcome: TOR (Time to Response)
Description: The time to achieve platelet count ≥ 50×10^9/L after switching.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
weeks | 5 [3 to 6] | 2 [1 to 4]

6. Secondary Outcome: DOR (Duration of Response)
Description: The duration of achieving platelet count ≥ 50×10^9/L after switching.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
Number analyzed (Participants) | 10 | 10
weeks | 3 [1 to 5] | 4 [1 to 5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Eltrombopag Group | Recombinant Human Thrombopoietin (Rh-TPO) Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag Group (N=10) | Recombinant Human Thrombopoietin (Rh-TPO) Group (N=10)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04214951/Prot_SAP_ICF_000.pdf